CLINICAL TRIAL: NCT04044170
Title: A Phase 2 Study of Poziotinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With EGFR or HER2 Exon 20 Mutation in China and Korea
Brief Title: Poziotinib in Patients With NSCLC Having EGFR or HER2 Exon 20 Insertion Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study termination by the Sponsor
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-PHI-202
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: NSCLC
MeSH Terms: interventions — HM781-36B

STUDY DESIGN:
Intervention Model Description: Each treatment cycle is 28 calendar days in duration. There will be two patient cohorts and eligible patients will be enrolled into each cohort in parallel based on EGFR or HER2 exon 20 mutation status:
  * Cohort 1 : Previously treated patients with EGFR exon 20 insertion mutation positive NSCLC
  * Cohort 2 : Previously treated patients with HER2 exon 20 insertion mutation positive NSCLC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poziotinib (Experimental): * Cohort 1 : Previously treated patients with EGFR exon 20 insertion mutation positive NSCLC
  * Cohort 2: Previously treated patients with HER2 exon 20 insertion mutation positive NSCLC
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
  Other Names: HM781-36B

SUMMARY:
This is a Phase 2, open-label, multicenter study to evaluate the efficacy and the safety/tolerability of poziotinib in two patient cohorts for up to 114 previously treated NSCLC patients with any systemic therapy (57 patients with EGFR exon 20 insertion mutations and 57 patients with HER2 exon 20 insertion mutations).

DETAILED DESCRIPTION:
The Screening period (Day -30 to Day -1) lasts up to approximately 30 days prior to Cycle 1, Day 1. Patients must meet all Inclusion/Exclusion Criteria to participate in the study. Eligible patients will provide written Informed Consent prior to any study procedures.

Each treatment cycle is 28 calendar days in duration. There will be two patient cohorts and eligible patients will be enrolled into each cohort in parallel based on EGFR or HER2 exon 20 mutation status:

* Cohort 1 : Previously treated patients with EGFR exon 20 insertion mutation positive NSCLC (N=57)
* Cohort 2 : Previously treated patients with HER2 exon 20 insertion mutation positive NSCLC (N=57) Toxicity will be assessed based on the severity grade of the adverse events using CTCAE version 4.03.

Poziotinib (16 mg) will be taken orally, once daily (QD) with food and a glass of water at approximately the same time each morning.

All patients will be treated until disease progression, death, intolerable adverse events (AEs), or other protocol-specified reasons for patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age (or country's legal age of majority if the legal age was > 18 years) at the time of obtaining informed consent.
2. Patient must be willing and capable of giving written Informed Consent, adhering to dosing and visit schedules, and meeting all study requirements
3. Patient has histologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) that is not amenable to treatment with curative intent
4. Patient has had at least one prior systemic treatment for NSCLC, but no more than three prior systemic therapy
5. Patient has adequate tumor tissue obtained from a biopsy or surgical procedure to enable molecular profiling for central laboratory confirmation of the mutation.
6. Patient is positive for EGFR or HER2 exon 20 mutations based on tissue testing:

   * Cohort 1: Documented EGFR exon 20 insertion mutation (including duplication mutations)
   * Cohort 2: Documented HER2 exon 20 insertion mutation (including duplication mutations)
7. Patient has measurable disease, as per the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1). Metastatic lesions in CNS or in brain cannot be used for target lesions.
8. Brain metastases may be allowed if patient's condition is stable.
9. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 and has a life-expectancy of more than 6 months
10. Patient has recovered from prior systemic therapy for metastatic disease to Grade ≤1 for non-hematologic toxicities (except for Grade ≤2 peripheral neuropathy) and has adequate hematologic, hepatic, and renal function at Baseline
11. Patient is willing to practice 2 forms of contraception, one of which must be a barrier method, from study entry until at least 30 days after the last dose of poziotinib
12. Females of childbearing potential must have a negative pregnancy test within 30 days prior to enrollment. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or who are surgically sterilized do not require this test.

Exclusion Criteria:

1. Patient has EGFR T790M mutation or any other acquired EGFR exon 20 point mutation
2. Patient has had previous treatment with poziotinib or any other EGFR or HER2 exon 20 insertion mutation-selective tyrosine kinase inhibitor (TKI) prior to study participation.
3. Patient has had radiotherapy (intention for cure) or surgery (other than surgical placement for vascular access and minimally invasive procedures including some biopsy procedures) within 2 weeks prior to start of study treatment with poziotinib
4. Patient has a history of congestive heart failure (CHF) Class III/IV according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment
5. Patient has a high risk of cardiac disease, as determined by the Investigator, may undergo either echocardiogram (ECHO) or multi-gated acquisition (MUGA) during Screening and has a cardiac ejection fraction <50%.
6. Patient has had other malignancies within the past 3 years, except for stable non-melanoma skin cancer, fully treated and stable early stage prostate cancer or carcinoma in situ of the cervix or breast without need of treatment
7. Patient is confirmed to have clinically significant or recent acute gastrointestinal disease presenting as diarrhea and/or coloenteritis as a main symptom.
8. Patient has an active Grade ≥2 skin disorder, rash, mucositis, or skin infection that needs medication or therapy or existing Grade ≥2 skin toxicity from previous therapies.
9. Presence or history of interstitial lung disease (ILD), drug-induced ILD, or presence of radiation pneumonitis
10. Patient is unable to take drugs orally due to disorders or diseases that may affect gastrointestinal function, such as inflammatory bowel diseases or malabsorption syndrome, or procedures that may affect gastrointestinal function
11. Patient has an active liver disease or biliary tract disease (except for Gilbert's disease, asymptomatic biliary stones, liver metastasis, or stabilized chronic liver diseases)
12. Patient has known hypersensitivity to poziotinib or has a history of allergic reactions attributed to chemically similar compounds or other tyrosine kinase inhibitors (TKIs)
13. Patient has an active uncontrolled infection, underlying medical condition, or other serious illness that would not be appropriate for this study
14. Patient has unstable, uncontrolled, active bleeding disorders that the investigator considers that the patient could be at increased risk or not be suitable for treatment in this study
15. Patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of poziotinib to the end of study.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  The proportion of subjects who achieve CR, PR, and Stable Disease (SD) by the best response from the first dose of poziotinib to the end of study.
Duration of Response (DoR) | 24 months
  Number of days from the date that measurement criteria are first met for CR or PR (whichever status is recorded first) until the first subsequent date that progressive disease or death is documented.
Progression-free Survival (PFS) | 24 months
  Number of days from the treatment start date to the date of documented disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Pharmaceuticals, Study Director — Hanmi Pharmaceuticals
Locations (26):
- China (21):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - Beijing Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Cancer Hospital and Institute, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Guangdong Panyu Central Hospital, Guangzhou
  - Shi Run Run Shaw Hospital, Zhejiang University, Hangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - Shanghai Chest Hospital, Shanghai
  - University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul